CLINICAL TRIAL: NCT05255497
Title: Effects of Balance Exercises in Diabetic Peripheral Neuropathy
Brief Title: The Effect of Sensorial Biodex Balance Balance System Exercises in Diabetic Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duygu AKTAR REYHANIOGLU (Other)
Responsible Party: Sponsor-Investigator, Duygu AKTAR REYHANIOGLU, Principal Investigator, Izmir Tinaztepe University
Organization: Izmir Tinaztepe University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: IzmirTinaztepeU
Record Dates: First submitted 2022-02-16; First posted 2022-02-24 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-02

CONDITIONS: Diabetic Neuropathies; Diabetes Mellitus; Exercise Training
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biodex Balance Group (Experimental): This group performed exercises using the biodex balance system
  Interventions: Device: Biodex Balance Exercise System
- Control Group (No Intervention): This group was informed about diabetes self-management.

INTERVENTIONS:
Device: Biodex Balance Exercise System — Patients in the intervention group (n=14) performed exercises using the computerized BBS. The control group (n=13) was just informed about diabetes self-management.
  Arms: Biodex Balance Group

SUMMARY:
This study examined the effects of balance exercises performed with the Biodex Balance System (BBS) on nerve conduction, sensory symptoms, and muscle strength in patients with diabetes-related neuropathy.

DETAILED DESCRIPTION:
We enrolled twenty-seven patients in this study. Patients in the intervention group (n=14) performed exercises using the computerized BBS. The control group (n=13) was just informed about diabetes self-management. All patients underwent pretest and posttest peripheral nerve conduction studies. Sensory examination performed by using 5.07 Semmes-Weinstein monofilaments and 128-Hz tuning fork. Muscle strength measurements obtained with manual dynamometer

ELIGIBILITY:
Inclusion Criteria:

* diabetes-related neuropathy based on laboratory tests, clinical findings, and nerve conduction study

Exclusion Criteria:

* increased risk of non-diabetes related neuropathy: history of autoimmune, cerebrovascular, or chronic infectious disease, cancer, chemotherapy and/or radiotherapy, radicular neuropathy, chronic kidney and liver failure, alcoholism or other substance abuse, and mental or physical disabilities (including blindness). We also excluded patients who didn't speak Turkish

Ages: 45 Years to 76 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-09-02 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2020-09-20 (Actual)

PRIMARY OUTCOMES:
The effect of biodex balance training on muscle strength was evaluated. | Change from baseline to 8 weeks
  Muscle test was evaluated with a manual dynamometer. The measurements of both groups before and after the training were compared.
The effect of biodex balance training on protective senses | Change from baseline to 8 weeks
  Protective senses was assessed with monofilament and 128 Hz tuning fork
The effect of biodex balance training on motor nerves | Change from baseline to 8 weeks
  Nerve conduction test was assessed with electromyograph

CONTACTS AND LOCATIONS:
Overall Officials: Gaye Yıldırım, Dr, Study Chair — Dokuz Eylul University
Locations (1):
- Dokuz Eylul University, Izmir, Balcova/Incialtı, Turkey (Türkiye)

REFERENCES:
- [Derived] Reyhanioglu DA, Yildirim G, Sengun IS, Kara B. Effects of Computer-based Balance Exercises on Balance, Pain, Clinical Presentation and Nerve Function in Patients With Diabetic Peripheral Neuropathy: A Randomized Controlled Study. J Musculoskelet Neuronal Interact. 2024 Jun 1;24(2):168-177. PMID 38825999